CLINICAL TRIAL: NCT02273388
Title: An Open Phase I Single Dose Escalation Study of BI 6727 Administered Intravenously in Patients With Advanced Solid Tumours With Repeated Administration in Patients With Clinical Benefit
Brief Title: BI 6727 Administered Intravenously Every 3 Weeks in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1230.1; 2005-002500-42 (EudraCT Number: EudraCT); 1230-0001 (Other: BI)
Record Dates: First submitted 2014-10-23; First posted 2014-10-24 (Estimated); Results first posted 2023-10-03 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2022-12

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — BI 6727

ARMS (12):
- 12 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 24 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 48 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 75 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 125 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 200 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 300 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 300 mg BI 6727 1h2h (Experimental): Infusion over 1 hour (1h) in course 1 and over 2 hours (2h) in course 2.
  Interventions: Drug: BI 6727
- 300 mg BI 6727 2h1h (Experimental): Infusion over 2 hours (2h) in course 1 and over 1 hours (1h) in course 2.
  Interventions: Drug: BI 6727
- 350 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 400 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727
- 450 mg BI 6727 (Experimental)
  Interventions: Drug: BI 6727

INTERVENTIONS:
Drug: BI 6727 — BI 6727
  Other Names: Volasertib

SUMMARY:
The primary objective of this trial is to identify the maximum tolerated dose (MTD) of BI 6727 therapy in terms of drug-related adverse events. Secondary objectives are the collection of overall safety and antitumour efficacy data and the determination of the pharmacokinetic profile of BI 6727.

ELIGIBILITY:
Inclusion criteria:

1. Patients with confirmed diagnosis of advanced, non resectable and / or metastatic solid tumours, who have failed conventional treatment, or for whom no therapy of proven efficacy exists, or who are not amenable to established forms of treatment
2. Age 18 years or older
3. Written informed consent consistent with ICH-GCP and local legislation
4. Eastern Cooperative Oncology Group (ECOG, R01-0787) performance score ¿ 2
5. Recovery from CTCAE Grade 2 - 4 therapy-related toxicities from previous chemo-, hormone-, immuno-, or radiotherapies (except alopecia)

   The 18 additional patients recruited at the MTD must also meet the following criterion:
6. Measurable tumour deposits (RECIST) by one or more techniques (CT, MRI)

Exclusion criteria:

1. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol
2. Pregnancy or breastfeeding
3. Active infectious disease or known chronic Hepatitis B/Hepatitis C infection
4. Clinical evidence of active brain or leptomeningeal disease during the past 12 months
5. Second malignancy currently requiring active therapy
6. Absolute neutrophil count less than 1500 / mm3
7. Platelet count less than 100 000 / mm3
8. Bilirubin greater than 1.5 mg / dl (> 26 ¿mol / L, SI unit equivalent)
9. Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
10. Serum creatinine greater than 1.5 mg / dl (> 132 ¿mol / L, SI unit equivalent)
11. Known history of relevant QT-prolongation, e.g. long QT-syndrome
12. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
13. Treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
14. Chemo-, radio or immunotherapy within the past four weeks before start of therapy or concomitantly with this trial. This restriction does not apply to steroids and bisphosphonates.
15. Patients unable to comply with the protocol
16. Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-11-04 (Actual); Primary Completion 2009-01-19 (Actual); Study Completion 2021-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Belgium (2):
  - 1230.1.32002 Boehringer Ingelheim Investigational Site, Brussels
  - 1230.1.32001 Boehringer Ingelheim Investigational Site, Leuven

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An open label, uncontrolled "first in man" dose escalation trial in patients with advanced solid tumours with repeated administration in patients with clinical benefit.
Pre-assignment Details: All patients were screened for eligibility to participate in the trial. Patients attended specialist sites to ensure that all patients met all inclusion/exclusion criteria. Patients were not to be entered to trial treatment if any one of the specific entry criteria were not met.
Groups:
- 12 mg BI 6727: 12 milligram (mg) solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 24 mg BI 6727: 24 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 48 mg BI 6727: 48 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 75 mg BI 6727: 75 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 125 mg BI 6727: 125 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 200 mg BI 6727: 200 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 300 mg BI 6727: 300 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 300 mg BI 6727 1h2h: 300 mg solution for injection of BI 6727 was administered as intravenous infusion over 1 hour (1h) in course 1 and over 2 hours (2h) in course 2 once every 21 days (as long as there was clinical benefit for the patients). QT extension cohort.
- 300 mg BI 6727 2h1h: 300 mg solution for injection of BI 6727 was administered as intravenous infusion over 2 hour (2h) in course 1 and over 1 hour (1h) in course 2 once every 21 days (as long as there was clinical benefit for the patients). QT extension cohort.
- 350 mg BI 6727: 350 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 400 mg BI 6727: 400 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
- 450 mg BI 6727: 450 mg solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients).
Period: Overall Study
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Started (Started are treated) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Adverse Event study disease worse | 4 | 3 | 3 | 2 | 4 | 3 | 14 | 6 | 6 | 5 | 10 | 1
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): The treated set consists of all patients who received at least one dose of BI 6727.
Groups:
- Total: Total of all reporting groups
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727 | Total
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2 | 65
Age, Continuous [Median (Full Range); unit: Years] | 34.5 [19 to 47] | 53.0 [43 to 62] | 43.0 [37 to 68] | 57.0 [51 to 63] | 58.5 [48 to 73] | 65.0 [59 to 71] | 55.0 [24 to 79] | 54.5 [41 to 66] | 60.5 [44 to 78] | 61.0 [57 to 79] | 60.0 [39 to 79] | 50.0 [41 to 59] | 58.0 [19 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 2 | 1 | 1 | 6 | 1 | 2 | 3 | 5 | 0 | 27
  Male | 1 | 0 | 3 | 0 | 3 | 2 | 9 | 7 | 4 | 2 | 5 | 2 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as: the dose of BI 6727 which is one dose tier below that dose at which two or more out of a maximum of six patients experienced dose-limiting toxicity (DLT). At the maximum tolerated dose, no more than one patient out of six patients may experience DLT, i.e. MTD is defined as the highest dose studied for which the incidence of dose-limiting toxicity is no more than 17% (i.e. 1/6 patients) during the first course.
  DLT is defined as drug related common terminology criteria for adverse events (CTCAE) grade 3 or 4 non haematological toxicity (except emesis or diarrhoea responding to supportive treatment), or drug related CTCAE grade 4 neutropenia for seven or more days and / or complicated by infection, or CTCAE Grade 4 thrombocytopenia .
Time Frame: 21 days (first treatment course).
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Number; unit: Milligram (mg)
Groups:
- BI 6727: Comprises all dose groups during the dose escalation phase. 12/24/48/75/125/200/300/350/400 and 450 milligram (mg) solution for injection of BI 6727 was administered as intravenous infusion over 60 minutes once every 21 days (as long as there was clinical benefit for the patients). 300 mg 1h2h solution for injection of BI 6727 was administered as intravenous infusion over 1 hour (1h) in course 1 and over 2 hours (2h) in course 2 once every 21 days (as long as there was clinical benefit for the patients). 300 mg 2h1h solution for infusion of BI 6727 was administered as intravenous infusion over 2 hour (2h) in course 1 and over 1 hour (1h) in course 2 once every 21 days (as long as there was clinical benefit for the patients).
Arm/Group | BI 6727
Number analyzed (Participants) | 65
Milligram (mg) | 400

2. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with adverse events. The events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v.3.0.
  Grade refers to the severity of adverse event. Grade 1: Mild AE; Grade 2: Moderate AE; Grade 3: Severe AE; Grade 4: Life-threatening or disabling AE; Grade 5: Death related to AE.
Time Frame: From first drug administration until last drug administration plus 21 days, up to 835 days.
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Participants
  Grade 1 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
  Grade 2 | 0 | 0 | 1 | 1 | 3 | 2 | 6 | 2 | 3 | 0 | 1 | 0
  Grade 3 | 1 | 1 | 0 | 0 | 1 | 0 | 4 | 3 | 2 | 2 | 2 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 6 | 2
  Grade 5 | 2 | 1 | 1 | 1 | 0 | 1 | 3 | 2 | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Clinically Relevant Abnormalities
Description: Number of participants with clinically relevant abnormalities, occurring in >5% of the total number of participants, is reported.
  Clinically relevant post baseline values with Common Terminology Criteria for Adverse Events (CTCAE) grades:
  * CTCAE grade ≥4 for White blood cell count (WBC) , Neutrophils (NEUT), NEUABS Lymphocytes (LMPH) if baseline CTCAE grade is not 4
  * CTCAE grade ≥3 for Haemoglobin (HGB), Platelets count (PLTCT), Alkaline phosphatase (ALKP), serum glutamic-oxaloacetic-transaminase (SGOT), serum glutamic pyruvic transaminase (SGPT), total bilirubin (TBILI), if baseline CTCAE grade is ≥3 increases of one grade
  * CTCAE grade ≥2 for other parameters, if baseline CTCAE grade is ≥2 increases of at least one grade
Time Frame: From baseline to the last value on treatment, up to 814 days.
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Participants
  Haematocrit | 1 | 2 | 1 | 1 | 2 | 3 | 10 | 4 | 2 | 4 | 7 | 1
  Haemoglobin | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 3 | 0
  Mean corpuscular volume (MCV) | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 2 | 1
  Platelets | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 4 | 2
  Red blood cell count (RBC) | 0 | 0 | 1 | 1 | 2 | 2 | 7 | 4 | 1 | 3 | 4 | 2
  White blood cell count (WBC) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 0
  Neutrophils | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 6 | 2
  Sodium | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0
  Alkaline phosphatase | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Lactate dehydrogenase (LDH) | 0 | 2 | 1 | 0 | 2 | 1 | 2 | 2 | 1 | 1 | 1 | 0
  Albumin | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 0 | 0 | 2 | 2 | 1
  Creatinine | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1
  Glucose | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 0 | 0 | 2 | 0

4. Secondary Outcome: Number of Participants With Change in Eastern Cooperative Oncology Group (ECOG) Patient Performance Score
Description: ECOG score: The scale of ECOG score is defined as a six point categorical scale as described ranging from 0 (asymptomatic) to 5 (death). ECOG score change from baseline to end of treatment is calculated, and defined as
  = ECOG score at end of treatment - ECOG score at baseline.
  Scale of ECOG score change:
  The ECOG score changes from baseline score are categorized on a three point categorical scale: Improved, unchanged, and deteriorated. Improvement or deterioration of performance status required a decrease or an increase from baseline, respectively, of at least one point on the ECOG scale. The number of patients per category ("improved", "unchanged", "deteriorated" "unknown") is reported.
Time Frame: At baseline and at end of treatment (up to 814 days).
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Participants
  Improved | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unchanged | 1 | 2 | 1 | 1 | 1 | 2 | 7 | 2 | 2 | 3 | 2 | 0
  Deteriorated | 2 | 1 | 2 | 1 | 3 | 1 | 7 | 5 | 4 | 2 | 8 | 2
  Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

5. Secondary Outcome: Electrocardiogram (ECG) - QTcF Change From Baseline
Description: Electrocardiogram (ECG) - QTcF change from baseline. QTcF intervals form the ECGs were analysed for changes during and after intravenous infusion of BI 300 mg dose over 1 hours and over 2 hours. For baseline ECG, the combined baseline, defined as the mean of the 2 triplicates at the time-point closest to but prior to the start of the infusion of both treatment courses, i.e. a common baseline is used for both treatment courses, was used. Mean is adjusted mean.
  Abbreviations:
  QTcF: QT interval, corrected for heart rate according to Fridericia's formula (seconds) = measured QT / (cube root of preceding RR interval) QT: Interval from the beginning of the Q wave to the end of the T wave on an ECG (seconds).
  CfB: Change from baseline.
Time Frame: At baseline and 5 minutes before infusion end, 1 hour after end of infusion and at 4 and 12 hours after start of infusion, at course 1.
Population: QT extension cohort: Patients treated with 300 mg BI6727 to investigate QTc changes, according to two different treatment schedules in course 1 and course 2, (300 mg BI 6727 1h2h and 300 mg BI 6727 2h1h). Results are reported for 300 mg over 1 hour infusion vs. 300 mg over 2 hours infusion. Only participants with non-missing data were included in the analysis.
Measure: Mean (90% Confidence Interval); unit: Millisecond (ms)
Groups:
- 300 mg BI 6727 1h: 300 mg solution for injection of BI 6727 was administered as intravenous infusion over 1 hour (1h). QT extension cohort.
- 300 mg BI 6727 2h: 300 mg solution for injection of BI 6727 was administered as intravenous infusion over 2 hours (2h). QT extension cohort.
Arm/Group | 300 mg BI 6727 1h | 300 mg BI 6727 2h
Number analyzed (Participants) | 13 | 11
Millisecond (ms)
  CfB to 5 minutes before infusion end | 17.79 [13.68 to 21.90] | 13.23 [8.83 to 17.64]
  CfB to 1 hours after infusion end | 13.99 [9.88 to 18.10] | 6.84 [2.44 to 11.25]
  CfB to 4 hours after infusion start | 10.65 [6.54 to 14.76] | 7.08 [2.67 to 11.48]
  CfB to 24 hours after infusion start | 4.33 [0.22 to 8.44] | -4.33 [-8.73 to 0.07]
Statistical Analysis 1: Comparison: 300 mg BI 6727 1h vs 300 mg BI 6727 2h; Change from baseline to 5 minutes before infusion end. Linear mixed model with sequence, course, treatment (both infusion types i.e. 1 hour duration and 2 hour duration) and time as fixed effects and treatment*time as interaction effect, as well as the continuous , fixed covariate of baseline value; Test type: Other; Difference of adjusted means = -4.56, 90% CI 2-sided [-10.59 to 1.48], Standard Error of Mean 3.61 — Comparison vs. 1 hour infusion [2h-1h]
Statistical Analysis 2: Comparison: 300 mg BI 6727 1h vs 300 mg BI 6727 2h; Change from baseline to 1 hour after infusion end. Linear mixed model with sequence, course, treatment (both infusion types i.e. 1 hour duration and 2 hour duration) and time as fixed effects and treatment*time as interaction effect, as well as the continuous , fixed covariate of baseline value; Test type: Other; Difference of adjusted means = -7.14, 90% CI 2-sided [-13.18 to -1.11], Standard Error of Mean 3.61 — Comparison vs. 1hour infusion [2h-1h]
Statistical Analysis 3: Comparison: 300 mg BI 6727 1h vs 300 mg BI 6727 2h; Change from baseline to 4 hours after infusion start. Linear mixed model with sequence, course, treatment (both infusion types i.e. 1 hour duration and 2 hour duration) and time as fixed effects and treatment*time as interaction effect, as well as the continuous , fixed covariate of baseline value; Test type: Other; Difference of adjusted means = -3.58, 90% CI 2-sided [-9.61 to 2.46], Standard Error of Mean 3.61 — Comparison vs. 1 hour infusion [2h-1h]
Statistical Analysis 4: Comparison: 300 mg BI 6727 1h vs 300 mg BI 6727 2h; Change from baseline to 24 hours after infusion start. Linear mixed model with sequence, course, treatment (both infusion types i.e. 1 hour duration and 2 hour duration) and time as fixed effects and treatment*time as interaction effect, as well as the continuous , fixed covariate of baseline value; Test type: Other; Difference of adjusted means = -8.66, 90% CI 2-sided [-14.70 to -2.63], Standard Error of Mean 3.61 — Comparison vs. 1 hour [2h-1h]

6. Secondary Outcome: Vital Signs - Blood Pressure
Description: Systolic blood pressure and diastolic blood pressure are reported.
Time Frame: At baseline.
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Median (Full Range); unit: Millimeter of mercury (mmHg)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Millimeter of mercury (mmHg)
  Systolic blood pressure | 126 [110 to 155] | 124 [107 to 148] | 124 [110 to 134] | 112 [100 to 124] | 110 [99 to 131] | 130 [116 to 164] | 125 [102 to 172] | 129 [100 to 146] | 148 [120 to 165] | 135 [110 to 149] | 144 [88 to 178] | 129 [128 to 130]
  Diastolic blood pressure | 74 [60 to 80] | 80 [68 to 90] | 78 [78 to 85] | 75 [70 to 80] | 71.5 [58 to 80] | 76 [72 to 90] | 80 [69 to 98] | 78.5 [67 to 89] | 86.5 [60 to 100] | 82 [70 to 90] | 81.5 [45 to 100] | 75 [70 to 80]

7. Secondary Outcome: Vital Signs - Pulse Rate
Description: Pulse rate is reported.
Time Frame: At baseline.
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Median (Full Range); unit: Beats per minute (bpm)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Beats per minute (bpm) | 88 [76 to 92] | 80 [72 to 98] | 88 [73 to 92] | 92 [88 to 96] | 91 [84 to 99] | 88 [66 to 96] | 78 [64 to 120] | 84 [59 to 97] | 75 [58 to 104] | 76 [67 to 100] | 82 [62 to 114] | 76 [74 to 78]

8. Secondary Outcome: Number of Participants With Unconfirmed Best Overall Response
Description: For solid tumours, evaluation of tumour response was assessed according to the Response Evaluation Criteria in Solid Tumours (RECIST) definition. The overall response of target and non-target lesions together with or without the appearance of new lesions as reported by the investigator was assessed on a four point categorical scale as complete response (CR), partial response (PR), stable disease (SD), and progressive disease (PD) according to the RECIST criteria. In order to best handle measurements that were non-evaluable (NEV) a modified version of the RECIST criteria was used. If a RECIST overall response was deemed NEV, it could be further classified into non-evaluable clinically progressive disease (NEVCPD ) or non-evaluable clinically non-progressive disease (NEVCNPD), depending on the subjective assessment of the investigator.
Time Frame: Up to 814 days.
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
  Stable disease | 1 | 2 | 1 | 0 | 1 | 1 | 7 | 4 | 2 | 1 | 5 | 1
  Non-evaluable, clinically non-progressive disease (NEVCNPD) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Progressive Disease (PD) or NEVCPD | 2 | 1 | 2 | 2 | 2 | 2 | 8 | 3 | 4 | 4 | 3 | 0
  Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Progression
Description: Number of participants with progression of disease.
  Progressive disease is defined according to the Response Evaluation Criteria in Solid Tumours (RECIST) as: At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter.
Time Frame: Up to 814 days.
Population: Treated Set (TS): All patients who received at least one dose of BI 6727.
Measure: Count of Participants; unit: Participants
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 4 | 3 | 15 | 8 | 6 | 5 | 10 | 2
Participants | 3 | 3 | 3 | 2 | 4 | 3 | 15 | 7 | 6 | 5 | 10 | 1

10. Secondary Outcome: Maximum Concentration of BI 6727 in Plasma (Cmax)
Description: Maximum concentration of BI 6727 in plasma (Cmax).
  Different time frame for dose groups 300 mg BI 6727 1h2h and 300 mg BI 6727 2h1h:
  For 300mg BI 6727 1h2h: At course 1: 0.083 hours before drug administration and at 1*, 2, 4, 8, 24 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
  For 300mg BI 6727 2h1h: At course 1: 0.083 hours before drug administration and at 1*, 2, 3, 4 and 24 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
Time Frame: At course 1: 0.083 hours before drug administration and at 0.25, 0.5, 075, 1*, 1.5, 2, 4, 8, 24, 48, 96, 168, 336 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
Population: Treated Set (TS): All patients who received at least one dose of BI 6727. Only patients with non-missing values were included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/ Milliliter (ng/mL)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 8 | 6 | 5 | 9 | 2
Nanogram/ Milliliter (ng/mL) | 18.8 (14.3) | 50.7 (12.4) | 91.1 (17.6) | 169.0 (11.7) | 234.0 (30.9) | 470.0 (57.6) | 758 (28.8) | 519.0 (60.3) | 246.0 (68.8) | 724.0 (23.6) | 1020.0 (20.9) | 1450.0 (8.81)

11. Secondary Outcome: Time From Dosing to Maximum Concentration (Tmax)
Description: Time from dosing to maximum concentration (tmax).
  Different time frame for dose groups 300 mg BI 6727 1h2h and 300 mg BI 6727 2h1h:
  For 300mg BI 6727 1h2h: At course 1: 0.083 hours before drug administration and at 1*, 2, 4, 8, 24 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
  For 300mg BI 6727 2h1h: At course 1: 0.083 hours before drug administration and at 1*, 2, 3, 4 and 24 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
Time Frame: as for outcome 10
Population: as for outcome 10
Measure: Median (Inter-Quartile Range); unit: Hours (h)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 8 | 6 | 5 | 9 | 2
Hours (h) | 0.667 [0.500 to 0.750] | 0.750 [0.750 to 1.25] | 0.500 [0.250 to 0.533] | 0.884 [0.767 to 1.00] | 0.533 [0.500 to 0.733] | 1.00 [0.500 to 1.03] | 0.750 [0.500 to 1.00] | 1.00 [0.967 to 1.01] | 2.00 [1.98 to 2.00] | 0.750 [0.750 to 0.867] | 0.750 [0.250 to 1.00] | 0.517 [0.250 to 0.783]

12. Secondary Outcome: Area Under the Concentration-time Curve of BI 6727 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of BI 6727 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf).
Time Frame: 0.083 hours before drug administration and at 0.25, 0.5, 075, 1*, 1.5, 2, 4, 8, 24, 48, 96, 168, 336 and 504 hours after start of infusion. (*Immediately prior to end of infusion of BI 6727).
Population: Only patients in the treated set who had non-missing values were included in the analysis. For arms with 0 patients analysed: No sufficient data had been collected to determine the terminal half-life T1/2, which is needed to analyse the PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram * Hours / Milliliter (ng*h/mL)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 0 | 0 | 5 | 9 | 2
Nanogram * Hours / Milliliter (ng*h/mL) | 149 (31.6) | 380 (38.9) | 778 (25.1) | 1270 (7.64) | 2140 (27.9) | 5670 (36.7) | 6540 (32.6) |  |  | 10000 (57.6) | 7510 (19.3) | 10900 (14.0)

13. Secondary Outcome: Area Under the Concentration-time Curve of BI 6727 in Plasma Over the Time Interval From 0 to the Last Quantifiable Time Point tz (AUC0-tz)
Description: Area under the concentration-time curve of BI 6727 in plasma over the time interval from 0 to the last quantifiable time point tz (AUC0-tz).
  Different time frame for dose groups 300 mg BI 6727 1h2h and 300 mg BI 6727 2h1h:
  For 300mg BI 6727 1h2h: At course 1: 0.083 hours before drug administration and at 1*, 2, 4, 8, 24 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
  For 300mg BI 6727 2h1h: At course 1: 0.083 hours before drug administration and at 1*, 2, 3, 4 and 24 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
Time Frame: 0.083 hours before drug administration and at 0.25, 0.5, 075, 1*, 1.5, 2, 4, 8, 24, 48, 96, 168, 336 and 504 hours after start of infusion (*immediately prior to end of infusion of BI 6727).
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram * Hours / Milliliter (ng*h/mL)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 8 | 6 | 5 | 9 | 2
Nanogram * Hours / Milliliter (ng*h/mL) | 101 (39.0) | 320 (52.0) | 636 (25.8) | 1110 (15.9) | 1800 (20.6) | 4780 (20.0) | 5680 (26.4) | 2420 (52.3) | 1730 (53.7) | 8230 (37.1) | 6990 (18.5) | 10300 (15.7)

14. Secondary Outcome: Terminal Rate Constant in Plasma (λz)
Description: Terminal rate constant in plasma (λz).
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1 / hour
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 0 | 0 | 5 | 9 | 2
1 / hour | 0.00715 (32.0) | 0.00649 (16.9) | 0.00446 (40.1) | 0.00552 (28.9) | 0.00454 (30.7) | 0.00464 (49.4) | 0.00658 (27.2) |  |  | 0.00582 (37.6) | 0.00784 (49.2) | 0.00688 (20.4)

15. Secondary Outcome: Terminal Half-life of the Analyte in Plasma (t1/2)
Description: Terminal half-life of the analyte in plasma (t1/2).
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 0 | 0 | 5 | 9 | 2
Hours (h) | 96.9 (32.0) | 107 (16.9) | 156 (40.1) | 126 (28.9) | 153 (30.7) | 149 (49.4) | 105 (27.2) |  |  | 119 (37.6) | 88.4 (49.2) | 101 (20.4)

16. Secondary Outcome: Mean Residence Time of BI 6727 in the Body After Intravenous Administration (MRT)
Description: Mean residence time of BI 6727 in the body after intravenous administration (MRT).
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours (h)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 0 | 0 | 5 | 9 | 2
Hours (h) | 113 (33.6) | 127 (11.3) | 174 (36.2) | 137 (40.4) | 164 (29.6) | 139 (74.1) | 99.5 (38.7) |  |  | 131 (62.4) | 82.5 (43.5) | 88.1 (5.99)

17. Secondary Outcome: Total Clearance of BI 6727 in the Plasma After Intravascular Adminstration (CL)
Description: Total clearance of BI 6727 in the plasma after intravascular adminstration (CL).
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter/Minute (mL/min)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 0 | 0 | 5 | 9 | 2
Milliliter/Minute (mL/min) | 1140 (32.2) | 876 (44.4) | 924 (20.2) | 918 (9.17) | 947 (23.4) | 547 (28.8) | 762 (32.6) |  |  | 583 (57.6) | 885 (19.4) | 689 (14.0)

18. Secondary Outcome: Apparent Volume of Distribution at Steady State Following Intravascular Administration (Vss)
Description: Apparent volume of distribution at steady state following intravascular administration (Vss).
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 0 | 0 | 5 | 9 | 2
Liter | 7730 (30.8) | 6670 (46.0) | 9630 (36.7) | 7520 (50.9) | 9320 (13.3) | 4580 (41.2) | 4450 (37.1) |  |  | 4570 (19.8) | 4380 (49.3) | 3640 (20.1)

19. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase λz Following an Intravascular Dose (Vz)
Description: Apparent volume of distribution during the terminal phase λz following an intravascular dose (Vz).
Time Frame: as for outcome 10
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 3 | 3 | 2 | 3 | 3 | 11 | 0 | 0 | 5 | 9 | 2
Liter (L) | 9530 (34.8) | 8100 (52.6) | 12400 (46.2) | 9980 (38.8) | 12500 (15.1) | 7070 (19.4) | 6940 (38.0) |  |  | 6010 (28.1) | 6770 (54.7) | 6000 (35.1)

20. Secondary Outcome: Amount of BI 6727 That is Eliminated in Urine From the Time Point 0 to Time Point 24 Hours (Ae0-24)
Description: Amount of BI 6727 that is eliminated in urine from the time point 0 to time point 24 hours (Ae0-24).
Time Frame: 5 minutes prior to the infusion on day 1, course 1 and up to 24 hours after the infusion.
Population: Only patients in the treated set (TS) who had non-missing values were included in the analysis. Descriptive statistics for the 200 mg group could not be evaluated, since plasma concentrations of BI 6727 was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram (µg)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 3 | 1 | 13 | 8 | 6 | 4 | 10 | 2
Microgram (µg) | 299 (12.4) | 493 (104) | 1580 (12.9) | 1170 (72.9) | 2120 (14.8) | NA (NA) — Descriptive statistics for the 200 mg group could not be evaluated, since plasma concentrations of BI 6727 was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 5960 (56.5) | 3280 (64.1) | 3800 (82.2) | 9790 (84.8) | 4820 (58.5) | 6010 (26.7)

21. Secondary Outcome: Amount of BI 6727 That is Eliminated in Urine From the Time Point 0 to Time Point 48 Hours (Ae0-48)
Description: Amount of BI 6727 that is eliminated in urine from the time point 0 to time point 48 hours (Ae0-48).
Time Frame: 5 minutes prior to the infusion on day 1, course 1 and up to 48 hours after the infusion.
Population: Only patients in the treated set (TS) who had non-missing values were included in the analysis. Descriptive statistics for 200mg and 350mg group could not be evaluated, since plasma concentrations of BI 6727 was only quantifiable in less than two-thirds of the patients, respectively. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram (µg)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 3 | 1 | 13 | 7 | 6 | 3 | 10 | 2
Microgram (µg) | 379 (26.1) | 618 (105) | 2030 (15.7) | 1380 (66.5) | 2630 (14.6) | NA (NA) — Descriptive statistics for the 200 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 7810 (58.8) | 4830 (76.7) | 5810 (81.6) | NA (NA) — Descriptive statistics for the 350 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 6650 (57.4) | 7930 (26.2)

22. Secondary Outcome: Fraction of BI 6727 Eliminated in Urine From Time Point 0 to Time Point 24 Hours (Fe0-24)
Description: Fraction of BI 6727 (percentage of dose) eliminated in urine from time point 0 to time point 24 hours (Fe0-24).
Time Frame: 5 minutes prior to the infusion on day 1, course 1 and up to 24 hours after the infusion.
Population: Only patients in the treated set (TS) who had non-missing values were included in the analysis. Descriptive statistics for 200 mg group could not be evaluated, since plasma concentrations of BI 6727 was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 3 | 2 | 3 | 2 | 3 | 1 | 13 | 8 | 6 | 4 | 10 | 2
Percentage of dose | 3.10 (12.1) | 2.38 (101) | 3.65 (12.8) | 1.67 (70.8) | 1.74 (13.1) | NA (NA) — Descriptive statistics for the 200 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 1.99 (56.0) | 1.09 (64.1) | 1.27 (82.2) | 2.80 (84.8) | 1.19 (58.4) | 1.42 (35.7)

23. Secondary Outcome: Fraction of BI 6727 Eliminated in Urine From Time Point 0 to Time Point 48 Hours (Fe0-48)
Description: Fraction of BI 6727 (percentage of dose) eliminated in urine from time point 0 to time point 48 hours (Fe0-48).
Time Frame: 5 minutes prior to the infusion on day 1, course 1 and up to 48 hours after the infusion.
Population: as for outcome 21
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of dose
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 3 | 1 | 13 | 7 | 6 | 3 | 10 | 2
Percentage of dose | 3.75 (27.0) | 2.98 (102) | 4.71 (16.2) | 1.98 (64.5) | 2.16 (11.1) | NA (NA) — Descriptive statistics for the 200 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 2.61 (58.3) | 1.61 (76.7) | 1.94 (81.6) | NA (NA) — Descriptive statistics for the 350 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 1.65 (57.2) | 1.87 (35.1)

24. Secondary Outcome: Renal Clearance of BI 6727 From the Time Point 0 to Time Point 24 Hours (CLr,0-24)
Description: Renal clearance of BI 6727 from the time point 0 to time point 24 hours (CLr,0-24).
Time Frame: 5 minutes prior to the infusion on day 1, course 1 and up to 24 hours after the infusion.
Population: as for outcome 22
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter/minutes (mL/min)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 3 | 1 | 11 | 6 | 4 | 4 | 9 | 2
Milliliter/minutes (mL/min) | 106 (11.5) | 87.6 (67.8) | 127 (11.8) | 48.4 (117) | 56.7 (11.4) | NA (NA) — Descriptive statistics for the 200 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 42.3 (69.3) | 34.5 (54.9) | 34.2 (58.3) | 66.7 (89.9) | 24.5 (82.9) | 21.6 (15.3)

25. Secondary Outcome: Renal Clearance of BI 6727 From the Time Point 0 to Time Point 48 Hours (CLr,0-48)
Description: Renal clearance of BI 6727 from the time point 0 to time point 48 hours (CLr,0-48).
Time Frame: 5 minutes prior to the infusion on day 1, course 1 and up to 48 hours after the infusion.
Population: Only patients in the treated set with non-missing values. For arms with 0 patients analysed: No sufficient data had been collected to determine the terminal half-life T1/2, which is needed to analyse the PK data. Descriptive statistics for 200 and 350 mg group could not be evaluated, since plasma concentrations of BI 6727 was only quantifiable in less than 2/3 of patients, respectively. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated as defined in TSAP.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter/minutes (mL/min)
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
Number analyzed (Participants) | 4 | 2 | 3 | 2 | 3 | 1 | 11 | 0 | 0 | 3 | 9 | 2
Milliliter/minutes (mL/min) | 99.8 (5.89) | 80.6 (62.2) | 118 (13.5) | 43.9 (116) | 51.6 (3.77) | NA (NA) — Descriptive statistics for the 200 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP) | 41.3 (71.8) |  |  | NA (NA) — Descriptive statistics for the 350 mg group could not be evaluated, since plasma concentrations was only quantifiable in less than two-thirds of the patients. Descriptive statistics is calculated in case that 2/3 patients of total could be evaluated, as defined in the trial statistical analysis plan (TSAP). | 25.8 (80.9) | 21.5 (14.6)

ADVERSE EVENTS:
Time Frame: From first drug administration until last drug administration plus 21 days, up to 835 days.
Description: Treated Set (TS): ALL patients who received at least one dose of BI 6727.
Arm/Group | 12 mg BI 6727 | 24 mg BI 6727 | 48 mg BI 6727 | 75 mg BI 6727 | 125 mg BI 6727 | 200 mg BI 6727 | 300 mg BI 6727 | 300 mg BI 6727 1h2h | 300 mg BI 6727 2h1h | 350 mg BI 6727 | 400 mg BI 6727 | 450 mg BI 6727
All-Cause Mortality (participants affected / at risk) | 3/4 | 2/3 | 1/3 | 1/2 | 1/4 | 1/3 | 6/15 | 4/8 | 2/6 | 0/5 | 2/10 | 0/2
Serious Adverse Events (participants affected / at risk) | 3/4 | 2/3 | 2/3 | 1/2 | 0/4 | 2/3 | 9/15 | 3/8 | 1/6 | 3/5 | 5/10 | 2/2
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 2/3 | 1/2 | 4/4 | 3/3 | 15/15 | 8/8 | 6/6 | 3/5 | 10/10 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 12 mg BI 6727 (N=4) | 24 mg BI 6727 (N=3) | 48 mg BI 6727 (N=3) | 75 mg BI 6727 (N=2) | 125 mg BI 6727 (N=4) | 200 mg BI 6727 (N=3) | 300 mg BI 6727 (N=15) | 300 mg BI 6727 1h2h (N=8) | 300 mg BI 6727 2h1h (N=6) | 350 mg BI 6727 (N=5) | 400 mg BI 6727 (N=10) | 450 mg BI 6727 (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fusobacterium infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral pericarditis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urogenital haemorrhage (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphadenectomy (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mesenteric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 12 mg BI 6727 (N=4) | 24 mg BI 6727 (N=3) | 48 mg BI 6727 (N=3) | 75 mg BI 6727 (N=2) | 125 mg BI 6727 (N=4) | 200 mg BI 6727 (N=3) | 300 mg BI 6727 (N=15) | 300 mg BI 6727 1h2h (N=8) | 300 mg BI 6727 2h1h (N=6) | 350 mg BI 6727 (N=5) | 400 mg BI 6727 (N=10) | 450 mg BI 6727 (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 7 | 1 | 0 | 2 | 8 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 1 | 2 | 4 | 2 | 4 | 2 | 3 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 0 | 1 | 3 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 2 | 1 | 4 | 0 | 2 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 1 | 3 | 3 | 7 | 5 | 5 | 1 | 5 | 2
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Obstruction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 2 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Neutropenic infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Blood urea decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2 | 0 | 1 | 3 | 2 | 1 | 2 | 2 | 1 | 3 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 0 | 1 | 0 | 2 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0 | 1 | 2 | 1 | 4 | 2 | 1 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Genital infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyuria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombosis in device (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2005-10-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT02273388/Prot_000.pdf
  • Statistical Analysis Plan (2009-08-07): https://cdn.clinicaltrials.gov/large-docs/88/NCT02273388/SAP_001.pdf